CLINICAL TRIAL: NCT01708096
Title: Mechanisms Behind Antidiabetic Effects by Gastric By-pass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Anders Thorell, Assoc. Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009/931-31/2
Record Dates: First submitted 2012-10-09; First posted 2012-10-16 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes Mellitus Typ 2 and Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modifast (Active Comparator): treated with VLD Modifast 1000 kcal/day in 2 weeks before gastric by-pass,
  Interventions: Dietary Supplement: Modifast
- Normal diet (Placebo Comparator): normal diet 2 weeks before gastric by-pass surgery
  Interventions: Dietary Supplement: Normal diet

INTERVENTIONS:
Dietary Supplement: Modifast — 2 weeks before gastric by-pass patients are treated with VLD, 1000 kcal/day
  Arms: Modifast
Dietary Supplement: Normal diet — normal diet 2 weeks before gastric by-pass
  Arms: Normal diet

SUMMARY:
The aim of the study is to develop new strategies in treatment of continuous increasing number of patients with type 2 diabetes by understanding how bariatric surgery cures or improves this condition.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes typ 2
* 18-70 years
* BMI > 35 kg/m2
* Treated with oral antidiabetic agents and/or insulin
* laparoscopic surgery

Exclusion Criteria:

* Pharmacological treatment (other then above) witch could affect glucose metabolism
* open surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 12-18 month after gastric bypass
  Insulin sensitivity measured by hyperinsulinemic normoglycemic clamp technique

SECONDARY OUTCOMES:
Weight reduction | 12-18 month after gastric bypass

OTHER OUTCOMES:
Insulin signaling and glucose transport in skeletal muscle | 12-18 month after gastric by-pass

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, Assoc Prof, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Stockholm, Stockholm County Council
  - Uppsala University Hospital, Uppsala